CLINICAL TRIAL: NCT05592223
Title: A Phase I Single Site Open Label Clinical Trial for the Development of a Human BCG Challenge Model to Assess TB Drugs and Vaccines.
Brief Title: Phase I Open Label BCG Clinical Trial Assessing TB Drugs and Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, James Kublin, Principal Staff, Scientist Vaccine and Infectious Disease Division, Fred Hutch, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10903; RG1122457 (Other: Fred Hutch)
Record Dates: First submitted 2022-10-13; First posted 2022-10-24 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- BCG Challenged-Isoniazid Treated (Active Comparator): Will receive INH in the dose of 300 mg for three days post BCG injection.
  Interventions: Drug: BCG Vaccine USP; Drug: Isoniazid
- BCG Challenged-Isoniazid Untreated (Placebo Comparator): Will not receive any INH or RIF dose.
  Interventions: Drug: BCG Vaccine USP
- BCG Challenged-RIF Treated (Active Comparator): Will receive RIF in the dose of 600 mg for seven days post BCG injection.
  Interventions: Drug: BCG Vaccine USP; Drug: Rifampin

INTERVENTIONS:
Drug: BCG Vaccine USP — 2x10^6 cfu Tice® BCG (ID)
  Other Names: BCG
Drug: Isoniazid — INH in the dose of 300 mg for three days post BCG injection.
  Other Names: INH
  Arms: BCG Challenged-Isoniazid Treated
Drug: Rifampin — RIF in the dose of 600 mg for seven days post BCG injection.
  Other Names: RIF
  Arms: BCG Challenged-RIF Treated

SUMMARY:
The purpose of the study is to develop a BCG challenge model for use in short term Phase I human trials capable of assessing the ability of TB drugs and/or vaccine-induced immune responses to impact in vivo mycobacterial replication as a method of assessing antimycobacterial agents and/or protective immunity elicited by vaccines or host-directed therapy. The trial will illuminate the nature of local and systemic immune responses to BCG and treatment response, as well as demonstrate our local capacity for newer, more innovative study designs.

DETAILED DESCRIPTION:
This is phase 1, open-label, randomized clinical protocol to develop a human challenge model using the licensed and available BCG VACCINE USP (TICE® strain) with and without INH or Rifampin (RIF). Part 1 will involve 10 participants who will be screened and consented, given an intradermal injection of BCG; five of these participants will receive oral INH for 3 days. Part 2 will involve 10 participants who will be screened and consented, given an intradermal injection of BCG; five of these participants will receive oral RIF for 7 days. All participants will undergo physical exams, clinical evaluations, blood draws, urine collections, skin biopsies, and pregnancy tests. This study will measure the rate of replication by utilizing qPCR and in vitro culture, systemic innate and adaptive immune responses, including humoral and cellular assay analyses and the evaluation and PPD/IGRA status.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to initiation of any study procedures,
* Are males or non-pregnant females between the ages of 18 and 45 years, inclusive,
* Women of childbearing potential in sexual relationships with men must use an acceptable method of preventing conception from 30 days prior to 3 months after Tice® BCG administration. Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy or successful device placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or < 1 year of the last menses if menopausal). Includes but is not limited to, sexual abstinence, monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject receiving Tice® BCG, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing ®, and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
* For women of childbearing potential, negative serum pregnancy test at screening and negative urine pregnancy test within 24 hours prior to enrollment and Tice® BCG administration,
* Are in good health, as judged by the investigator and determined by vital signs (oral temperature, pulse, and blood pressure), medical history and physical examination,
* Have a negative HIV-1 ELISA test,
* Have negative serology tests for hepatitis B surface antigen and hepatitis C virus antibody,
* Have a negative QuantiFERON-TB Gold test,
* Negative is defined as Nil response < 0.8 IU/ml and TB Antigen response minus Nil response <0.35 IU/mL or TB Antigen response minus Nil response > 0.35 IU/mL and < 25% of Nil response and Mitogen response minus Nil response > 0.5 IU/ml,
* Have a urine dipstick for protein less than 1,
* Have a urine dipstick negative for glucose,
* Ability to understand and complete all study visits as required per protocol and be reachable by telephone.

Exclusion Criteria:

* Have a history of suspected, confirmed, treated or have other evidence of active tuberculosis,
* Symptoms may include recurrent fever, fatigue, night sweats, weight loss, oral ulcers, diarrhea, nausea, vomiting, or bleeding,
* Have any systemic symptoms* within 72 hours before Tice® BCG administration or signs of lymphadenopathy, hepatosplenomegaly, or pulmonary disease by physical examination on day of Tice® BCG administration. Includes fever, chills, malaise, fatigue, headache, night sweats, weight loss, nausea, vomiting, bleeding, diarrhea, abdominal pain, rhinorrhea, cough, wheezing, or shortness of breath.
* Have history of any significant acute or chronic medical conditions* or need for chronic medications that, in the opinion of the investigator, will interfere with immunity or affect safety. Includes, but is not limited to, disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic or autoimmune/inflammatory conditions. Have any history of excessive scarring or keloid formation.
* Have household contact or occupation involving significant contact with someone who is immunocompromised. Includes persons with HIV, AIDs, or active cancer; infants (children < 1 year); pregnant women; or persons who are immunosuppressed for approximately 6 weeks (during the time of active ID lesion drainage).
* Have a history of epilepsy (does not include febrile seizures as a child),
* Have a pacemaker, prosthetic valve, or implantable cardiac devices,
* Have a history of bleeding disorder,
* Have a known allergy to any Tice® BCG components (glycerin, asparagine, citric acid, potassium phosphate, magnesium sulfate, iron ammonium citrate, and lactose),
* Received blood products or immunoglobulin within 6 months prior to Tice® BCG administration,
* Received immunotherapy within one year prior to Tice® BCG administration,
* Received or plan to receive live attenuated vaccines 4 weeks before or after Tice® BCG administration,
* Received or plan to receive inactivated or killed vaccines 2 weeks before or after Tice® BCG administration,
* Plans to enroll in another clinical trial* that could interfere with safety assessment of the investigational product at any time during the study period. Includes trials that have a study intervention such as a drug, biologic, or device.
* Received an experimental agent* within 30 days prior to Tice® BCG administration or planned receipt of an experimental agent within 90 days after Tice® BCG administration, Includes vaccine, drug, biologic, device, blood product, or medication.
* Have a history of use of a systemic antibiotic within 14 days prior to Tice® BCG administration or planned use of a systemic antibiotic for 3 months after Tice® BCG administration,
* Have any medical, psychiatric, occupational, or behavioral problems that make it unlikely for the subject to comply with the protocol as determined by the investigator,
* Are health care providers at the highest risk of acquiring MTB infection, such as pulmonologists performing bronchoscopies on TB patients,
* Are breastfeeding or plan to breastfeed at any given time throughout the study,
* Have long term use of high dose oral or parenteral glucocorticoids, or high-dose inhaled steroids. Defined as taken for 2 weeks or more in total at any time during the past 2 months. High dose defined as prednisone ≥ 20 mg total daily dose, or equivalent dose of other glucocorticoids. High dose defined as > 800 mcg/day of beclomethasone dipropionate or equivalent. If short term corticosteroids are given, then the subject should not receive Tice® BCG or have blood collected for immunogenicity studies within 1 week of steroid administration.
* Have immunosuppression or are taking systemic immunosuppressants as a result of an underlying illness or treatment,
* Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 36 months prior to Tice® BCG administration,
* Any active neoplastic disease,
* Have a pulse rate less than 50 bpm or greater than 100 bpm,
* Have a systolic blood pressure less than 90 mm Hg or greater than 140 mm Hg,
* Have a diastolic blood pressure less than 50 mm Hg or greater than 90 mmHg,
* Have a WBC less than 4.0x103/uL or greater than 10.5x103/uL,
* Have hemoglobin less than 11.5x103/uL (female) or less than 12.5x103/uL (male),
* Have a platelet count less than 140x103/UL,
* Have a creatinine greater than 1.30 mg/dL,
* Have an ALT (SGPT) greater than 40 IU/L (female) or greater than 55 IU/L (male),
* Have known HIV, Hepatitis B, or Hepatitis C infection,
* Have a history of alcohol or drug abuse in the last 5 years,
* Have had a positive PPD skin test in the past or received BCG vaccine (BCG vaccination history will be determined by self-report, country of birth, and/or evidence of BCG scar),
* Have a BMI >35,
* PPD skin test within 2 months prior to Tice® BCG administration or planned receipt during the study other than from participation in this study,
* Oral temperature ≥ 100.4°F (≥ 38.0°C) or other symptoms of an acute illness within 3 days before Tice® BCG administration. (Subject may be rescheduled),
* Any medical disease or condition that, in the opinion of the investigator, is a contraindication to study participation. Includes medical disease or condition that would place the subject at an unacceptable risk of injury, render them unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or their successful completion of the study.
* Have any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol or compromise the interpretation of data or the scientific integrity of the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Kublin, MD, MPH, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing de-identified AE's/SAE's from all individual participants with Merck & Co during the trial.
Supporting Information: Study Protocol, ICF
Time Frame: During the participants active study period.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort A recruitment period 01 NOV 2022-01 DEC 2022 Cohort B recruitment period 01 JUL 2023-01 AUG 2023
Groups:
- BCG Challenged-Isoniazid Treated: Received INH at a dose of 300 mg for three days post BCG injection.
  BCG Vaccine USP: 2x10^6 cfu Tice® BCG (ID)
  Isoniazid: INH in the dose of 300 mg for three days post BCG injection.
- BCG Challenged-Isoniazid Untreated: Did not receive any INH dose.
  BCG Vaccine USP: 2x10^6 cfu Tice® BCG (ID)
- BCG Challenged-RIF Treated: Did receive RIF in the dose of 600 mg for seven days post BCG injection.
  BCG Vaccine USP: 2x10^6 cfu Tice® BCG (ID)
  Rifampin: RIF in the dose of 600 mg for seven days post BCG injection.
- BCG Challenged-Rifampin Untreated: Did not receive any Rif dose.
  BCG Vaccine USP: 2x10^6 cfu Tice® BCG (ID)
Period: Overall Study
Arm/Group | BCG Challenged-Isoniazid Treated | BCG Challenged-Isoniazid Untreated | BCG Challenged-RIF Treated | BCG Challenged-Rifampin Untreated
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCG Challenged-Isoniazid Treated | BCG Challenged-Isoniazid Untreated | BCG Challenged-RIF Treated | BCG Challenged-Rifampin Untreated | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Customized [Median (Full Range); unit: years]
  Median Age (Range) | 28 [20 to 36] | 40 [29 to 43] | 31 [21 to 41] | 36 [24 to 45] | 35 [20 to 45]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 3 | 3 | 2 | 3 | 11
  Female | 2 | 1 | 3 | 2 | 8
  Intersex | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 1 | 4
  Not Hispanic or Latino | 4 | 5 | 3 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 4 | 4 | 0 | 4 | 12
  More than one race | 1 | 0 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Assess Viable BCG Bacteria From Intradermal Challenge Site From Culture.
Description: Through microbial culture, quantify in colony forming units (CFU) BCG bacterial burden in skin biopsies from challenge sites. Outcome measure if the mean cfu from day 15 biopsy specimens.
Time Frame: 15 days after BCG dosing
Measure: Mean (Standard Deviation); unit: CFU
Arm/Group | BCG Challenged-Isoniazid Treated | BCG Challenged-Isoniazid Untreated | BCG Challenged-RIF Treated | BCG Challenged-Rifampin Untreated
Number analyzed (Participants) | 5 | 5 | 5 | 5
CFU | 20,440 (40,516) | 80 (92) | 5 (12) | 10,673 (12,646)

2. Secondary Outcome: The Rate of AE's/SAE's
Description: Mild (grade 1): events do not require treatment and do not interfere with the patient's daily activities
  Moderate (grade 2): events result in a low level of inconvenience or concern with the therapeutic measures. Moderate events may cause some interference with functioning and daily activities
  Severe (grade 3): events interrupt a patient's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually incapacitating.
Time Frame: Through study completion, an average of 16 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | BCG Challenged-Isoniazid Treated | BCG Challenged-Isoniazid Untreated | BCG Challenged-RIF Treated | BCG Challenged-Rifampin Untreated
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants
  All AEs: Number experiencing any Adverse Event | 5 | 4 | 4 | 5
  All AEs: Number experiencing no Adverse Events | 0 | 1 | 1 | 0
  Grade 3 AEs: Number experiencing any Adverse Event | 0 | 1 | 0 | 0
  Grade 3 AEs: Number experiencing no Adverse Events | 5 | 4 | 5 | 5

3. Secondary Outcome: Assess Quantitative Bacterial 16S Ribosomal DNA PCR
Description: Assessing the number of real time BCG genomes present in skin biopsies from challenge sites.
Time Frame: Day 15 post BCG dosing
Population: One participant declined day 15 biopsy
Measure: Mean (Standard Deviation); unit: copies
Arm/Group | BCG Challenged-Isoniazid Treated | BCG Challenged-Isoniazid Untreated | BCG Challenged-RIF Treated | BCG Challenged-Rifampin Untreated
Number analyzed (Participants) | 5 | 4 | 5 | 5
copies | 8239.4 (15243.9) | 97.7 (115.9) | 5.34 (11.9) | 10,673.4 (12645.7)

4. Secondary Outcome: Quantification by AUC of IgG in the Blood After BCG Immunization and INH or RIF Dosing.
Description: To assess the IgG immune response after INH or RIF dosing. The AUC we report is not a integration of concentration over time. Instead, AUC reported here quantifies the overall antibody binding signal across a titration series from a single time point (Day 144). In this assay, each sample from a single visit is measured at multiple dilutions, and the signal is expressed AUC in unit MFI × log₁₀(dilution). Plotting MFI as a function of dilution generates a curve that reflects how strongly and consistently the antibodies bind over the dilution range. The AUC therefore summarizes the entire binding titration curve - capturing both signal intensity and how long the signal is maintained across dilutions.
Time Frame: Day 144
Measure: Median (95% Confidence Interval); unit: MFI × log₁₀ dilution
Arm/Group | BCG Challenged-Isoniazid Treated | BCG Challenged-Isoniazid Untreated | BCG Challenged-RIF Treated | BCG Challenged-Rifampin Untreated
Number analyzed (Participants) | 5 | 5 | 5 | 5
MFI × log₁₀ dilution | 319.4 [276.3 to 469.1] | 822.5 [192.0 to 946.3] | 2888.8 [1941.878 to 4600.566] | 1951.5 [888.232 to 3436.136]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected through day 114 after vaccination
Arm/Group | BCG Challenged-Isoniazid Treated | BCG Challenged-Isoniazid Untreated | BCG Challenged-RIF Treated | BCG Challenged-Rifampin Untreated
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG Challenged-Isoniazid Treated (N=5) | BCG Challenged-Isoniazid Untreated (N=5) | BCG Challenged-RIF Treated (N=5) | BCG Challenged-Rifampin Untreated (N=5)
Severe Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — On Day 3 after vaccination participant suffered a severe back spasm and required treatment in the emergency department. Full function was regained and the SAE was considered non-study related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG Challenged-Isoniazid Treated (N=5) | BCG Challenged-Isoniazid Untreated (N=5) | BCG Challenged-RIF Treated (N=5) | BCG Challenged-Rifampin Untreated (N=5)
BCG Site Abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — One participant developed a sustained granulomatous fluid collection at the site of BCG injection. He required drainage and treatment with isoniazid. resolved 8 months after BCG injection.
Injection site erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 5 (5) | 5 (5)
Injection Site induration (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT05592223/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05592223/ICF_000.pdf